CLINICAL TRIAL: NCT04718142
Title: Variable Negative External Pressure (vNEP) - An Alternative to Continuous Positive Airway Pressure (CPAP) for the Treatment of Obstructive Sleep Apnea (OSA): A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somne, LLC (Industry)
Collaborators: California Center for Sleep Disorders (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20193101
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: negative pressure; variable negative external pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- vNEP with various shapes and sizes and overnight PSG (Experimental): Administer vNEP therapy to study participants on the throat's anterior surface with a variable negative pressure ranging from -20 cmH2O up to -35 cmH2O. Assess participants for a reduction in Apnea-Hypopnea Index (AHI) for at least 120 minutes using polysomnography (PSG) and treatment tolerance compared to CPAP.
  Interventions: Device: vNEP

INTERVENTIONS:
Device: vNEP — Apply vNEP therapy to the anterior surface of the throat with a variable negative pressure ranging from -20 cmH2O up to -35 cmH2O and vNEP devices of varying shapes and sizes.

SUMMARY:
Non-compliance rates estimated at 50% pose a major issue for CPAP therapy, the primary treatment for OSA. Negative external pressure, applied over the anterior neck under the mandible, has shown encouraging results as an alternative therapy. This study assessed a variety of sizes and shapes of collars and a range of pressures for variable negative external pressure (vNEP) treatment in subjects having moderate OSA to identify combinations that improve the efficacy and comfort of this emerging therapy.

Observations made in this study may be used to plan a more definitive follow-on investigation.

ELIGIBILITY:
Inclusion Criteria:

* a polysomnogram study or home sleep test within the previous six months that shows either an AHI > 15 and AHI <= 30
* able, in the opinion of the investigator, to understand and comply with all study procedures
* the vNEP collar is determined by the investigator to properly fit the subject and is well-tolerated after application to the neck.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Complete response | For 120 min
  Decrease in AHI <=5
Response | For 120 min
  Decrease in AHI of >=50% from baseline

SECONDARY OUTCOMES:
No response | For 120 min
  Did not achieve Primary Outcome Measure

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Kram, MD, Principal Investigator — California Center for Sleep Disorders
Locations (1):
- California Center for Sleep Disorders, San Leandro, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SA, Amis TC, Byth K, Larcos G, Kairaitis K, Robinson TD, Wheatley JR. Heavy snoring as a cause of carotid artery atherosclerosis. Sleep. 2008 Sep;31(9):1207-13. PMID 18788645
- [Background] Friedman M, Shnowske K, Hamilton C, Samuelson CG, Hirsch M, Pott TR, Yalamanchali S. Mandibular advancement for obstructive sleep apnea: relating outcomes to anatomy. JAMA Otolaryngol Head Neck Surg. 2014 Jan;140(1):46-51. doi: 10.1001/jamaoto.2013.5746. PMID 24263288
- [Background] Gelardi M, Del Giudice AM, Cariti F, Cassano M, Farras AC, Fiorella ML, Cassano P. Acoustic pharyngometry: clinical and instrumental correlations in sleep disorders. Braz J Otorhinolaryngol. 2007 Mar-Apr;73(2):257-65. doi: 10.1016/s1808-8694(15)31075-2. PMID 17589736
- [Background] Kais SS, Klein KB, Rose RM, Endemann S, Coyle WJ. Continuous negative external pressure (cNEP) reduces respiratory impairment during screening colonoscopy: a pilot study. Endoscopy. 2016 Jun;48(6):584-7. doi: 10.1055/s-0042-102533. Epub 2016 Apr 25. PMID 27110692
- [Background] Kendzerska T, Grewal M, Ryan CM. Utility of Acoustic Pharyngometry for the Diagnosis of Obstructive Sleep Apnea. Ann Am Thorac Soc. 2016 Nov;13(11):2019-2026. doi: 10.1513/AnnalsATS.201601-056OC. PMID 27529798
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Derived] Kram JA, Pelayo R. Variable negative external pressure-an alternative to continuous positive airway pressure for the treatment of obstructive sleep apnea: a pilot study. J Clin Sleep Med. 2022 Jan 1;18(1):305-314. doi: 10.5664/jcsm.9680. PMID 34596039
- See also: Rose RM, Aarestad J, Flicker W et al. Effect of continuous negative external pressure (cNEP) on upper airway (UA) structure and function: implications for obstructive sleep apnea and anesthesia care. Presented at the annual meeting of the America Society — http://www.asaabstracts.com/strands/asaabstracts/abstract.htm?year=2011&index=18&absnum=7646